CLINICAL TRIAL: NCT01453062
Title: Phase IV Observational Study in Chronic Lymphocytic Leukemia Patients Receiving Ofatumumab in the European Union
Brief Title: Phase IV Observational Study in Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114429; WEUSRTP4799 (Other: GSK); EPI40635 (Other: GSK)
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: Ofatumumab; Chronic lymphocytic leukemia (CLL); Arzerra
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of CLL: Patients with a diagnosis of CLL
  Interventions: Drug: Arzerra

INTERVENTIONS:
Drug: Arzerra — Treatment with Arzerra

SUMMARY:
B-cell chronic lymphocytic leukemia (CLL) is a subtype of mature peripheral B-cell neoplasms, characterized by the accumulation of circulating malignant lymphocytes that typically express cell surface markers CD5, CD20, and CD23. It is the most common type of leukemia in adults in Western Europe and in the US. The median age at diagnosis is 65-70 years, with a male to female ratio of 2:1. Initially, most patients present with asymptomatic lymphocytosis and do not need cytoreductive therapy. Patients with active disease are characterized by a lymphocyte doubling time of less than 6 months, or progressive, even massive lymphadenopathy, hepatosplenomegaly, anemia and thrombocytopenia. Constitutional symptoms such as fever, night sweats, unintended weight loss, and extreme fatigue are common in advanced disease and can significantly impact quality of life. CLL also causes relative immunosuppression that increases the risk of infections that are ultimately the major cause of death in this patient population. Median survival at diagnosis ranges from 5 to 20+ years depending on risk factors, but is only 6 to 14 months for patients with CLL refractory to available therapies.

Arzerra (ofatumumab) is a human monoclonal antibody (IgG1) that binds specifically to a distinct epitope encompassing both the small and large extracellular loops of the CD20 molecule. The CD20 molecule is a transmembrane phosphoprotein expressed on B lymphocytes from the pre-B to mature B lymphocyte stage and on B-cell tumors.

Arzerra is designated as an orphan medicinal product in the European Union (EU) for treatment of chronic lymphocytic leukemia. The Committee for Orphan Medicinal Products (COMP) concluded that chronic lymphocytic leukemia was estimated to be affecting approximately 3.5 in 10,000 persons in the Community at the time the application was made (June 2008) and that the condition is chronically debilitating and life-threatening, in particular due to poor long-term survival in high-risk patients.

Arzerra was given a conditional approval in the EU on April 19, 2010. The approved indication in the EU for the product is treatment of CLL in patients refractory to fludarabine and alemtuzumab. A specific obligation for this conditional approval was an agreement by GSK to conduct a post-marketing observational study in CLL patients receiving Arzerra. The data from this study is intended to enhance the evidence of the safety and efficacy of Arzerra as it is used in clinical practice, and once final data are available, together with results of a second specific obligation study, will support the transition from conditional to a full approval of Arzerra in the EU.

The objective of this observational study is to provide additional data to confirm the safety profile and efficacy of Arzerra for CLL patients treated in clinical practice.

Particular data of interest are: co-morbidities (specific chronic disease diagnoses), concomitant medications, disease (CLL) characteristics, prior treatment regimens, adverse events, reasons for discontinuation of Arzerra therapy, Arzerra response, progression free survival, and overall survival.

This is an observational, non-interventional, medical record review study in CLL patients. A total of 100 patients with CLL who have previously received Arzerra, whether alive or deceased, and have either completed the full course of Arzerra therapy or discontinued treatment early will be eligible to participate in the study. Centers across Europe who are members and non members of the European Research Initiative of CLL (ERIC) and treat CLL patients will participate in the study.

CLL patients newly initiating Arzerra who are still undergoing the treatment phase and patients having been treated with Arzerra in phase II or phase III clinical trials will be excluded.

For patients who have completed approximately 1 year or more of follow up since Arzerra initiation, data on response to Arzerra, adverse events during treatment and subsequent to treatment, patient status, progression free survival and overall survival covering the period up to approximately one-year post-drug initiation will be collected. For patients who have not completed approximately l year of follow-up since Arzerra initiation, including those who have been lost to follow up or died prior to one year or have not yet had a full year to elapse in calendar time, similar data will be collected at the point in time at the last available patient contact with the physician using information in the record. After approach for informed consent from the patient or next of kin for patients who have died to review the medical record, no interaction with the patient will occur.

ELIGIBILITY:
Inclusion Criteria:

* All CLL patients who have previously received Arzerra, whether alive or deceased
* Patients who have either completed the full course of Arzerra therapy or discontinued treatment early

Exclusion Criteria:

* CLL patients newly initiating Arzerra
* Patients having been treated with Arzerra in phase II or phase III clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 100 patients with CLL who have previously received Arzerra, whether alive or deceased, and have either completed the full course of Arzerra therapy or discontinued treatment early.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Physicians' assessment of response | Approximately one-year post-drug initiation or at the last available patient contact with the physician
  Physicians' assessment of response to include one or more of the following: CR, MRD status, incomplete CR, PR nodular, Stable Disease, Refractory/Progressive disease

SECONDARY OUTCOMES:
Adverse events | Approximately one-year post-drug initiation or at the last available patient contact with the physician
Progression-free survival | Approximately one-year post-drug initiation or at the last available patient contact with the physician
Overall survival | Approximately one-year post-drug initiation or at the last available patient contact with the physician

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Moreno C, Montillo M, Panayiotidis P, Dimou M, Bloor A, Dupuis J, Schuh A, Norin S, Geisler C, Hillmen P, Doubek M, Trneny M, Obrtlikova P, Laurenti L, Stilgenbauer S, Smolej L, Ghia P, Cymbalista F, Jaeger U, Stamatopoulos K, Stavroyianni N, Carrington P, Zouabi H, Leblond V, Gomez-Garcia JC, Rubio M, Marasca R, Musuraca G, Rigacci L, Farina L, Paolini R, Pospisilova S, Kimby E, Bradley C, Montserrat E. Ofatumumab in poor-prognosis chronic lymphocytic leukemia: a phase IV, non-interventional, observational study from the European Research Initiative on Chronic Lymphocytic Leukemia. Haematologica. 2015 Apr;100(4):511-6. doi: 10.3324/haematol.2014.118158. Epub 2015 Jan 16. PMID 25596264